CLINICAL TRIAL: NCT03404583
Title: Person-centred eHealth for Treatment and Rehabilitation of Severe Stress and Burnout Syndrome - a Randomized Controlled Trial in Primary Health Care
Brief Title: Person-centred eHealth for Treatment and Rehabilitation of Severe Stress and Burnout Syndrome
Acronym: PROMISE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Göteborg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PROMISE
Record Dates: First submitted 2018-01-12; First posted 2018-01-19 (Actual); Last update posted 2020-08-27 (Actual); Status verified 2020-08

CONDITIONS: Mental Health
Keywords: Person-centred care
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Person-centred care at distance (Experimental): Person-centred care at distance through an eHealth platform
  Interventions: Behavioral: Person-centred care at distance through an eHealth platform
- Usual Care (No Intervention): Evidence-based care

INTERVENTIONS:
Behavioral: Person-centred care at distance through an eHealth platform — Person-centred care at distance through an eHealth platform, used by professionals, patients and relatives
  Arms: Person-centred care at distance

SUMMARY:
The goal of the research project PROMISE is to translate the person-centred care (PCC) principles into an eHealth (the use of information and communication technologies for health) context. A developed PCC eHealth platform will be used as a tool to identify patients´ resources to enhance coping and living with their illness by means of a dialog and partnership with staff and relatives. The PCC eHealth platform will not replace, but instead be used as add on treatment to usual care (guideline directed care).

DETAILED DESCRIPTION:
A pilot study and collaboration between patients, relatives and professionals in the research program has clarified the need to develop a PCC eHealth platform. Previous research has shown that eHealth support, where the users are not involved in the process, has a low impact and has highlighted several limitations with respect to: patients' participation in the design process; its anchorage in the home and local environment and opportunities for communication rather than information. Therefore this study has a participatory design which assumes that all users (patients, relatives and health care professionals) are involved in the study design which facilitates implementation. An end-user perspective as a starting point increases the chances that users adapt a positive attitude towards the new system. Person-centred care combined with an eHealth support along the chain of health care showed a 4-fold chance of improved self-efficacy in combination with return to work or prior activity level after an event of acute coronary syndrome.

The aim of this project is that PCC can be delivered at distance and make health care more effective above and beyond usual care. Inclusion of the principles of PCC in an eHealth support for patients with stress, depression or anxiety will improve return to work rates, reduced relapse, reduce costs and improved self-efficacy.

In the PCC approach, the aims, capabilities and needs of each patient, will be the starting point. Self-care strategies will be reinforced and empowered.

This study is a randomized, open, parallel group intervention study where patients are eligible when they start their sick leave period due to stress, depression or anxiety. They will be asked about participation after being diagnosed and their sick leave has been approved.

Patients will be randomized into either the control or the intervention arm 1:1. The control group will receive usual care. The intervention group will receive usual care plus a PCC intervention through an eHealth platform. Randomization will be done through computer generated lists and stored in sealed envelopes.

Patients listed in primary care with a confirmed diagnosis of stress, depression or anxiety will be screened and sent an informing letter about the study from the chief at each centre. Specially trained registered nurses (RNs) will then screen patients against study inclusion and exclusion criteria and by phone contact eligible patients and inform the patient about the aims of the study and ask if they are interested to participate. If the patient wants to participate a consent form is sent to the patient and then returned to the RN. Written informed consent will then be obtained. Then the randomization procedure is performed which is stratified for age (≥ 50y) and diagnosis (stress, depression and anxiety) and the patient will be informed about the outcome by phone. Patients randomized to the intervention group will need a computer, smart phone or iPad to participate in the study.

Two dedicated full-time RNs follow the procedures closely. A monitor controls the protocol adherence. All case record forms, questionnaires and referrals will be constructed (for intervention and usual care groups).

Follow-up questionnaires on general self-efficacy, self-efficacy (self-care) quality of life, anxiety and depression, symptom burden and daily functional level will be sent out to all patients in both groups after 3,6,12,18 and 24 months after randomization.

Patients randomized to usual care will be managed by regular evidence-based treatment and care as outlined in treatment guidelines and followed as usual at their local primary care centre.

Patients will be contacted by a RN who has received special training in PCC communication at distance through the eHealth platform, for an initial person-centred dialogue by phone. Based on the patient narrative patient´s goals, resources and needs are identified. The patient (sometimes maybe together with relatives) and the RN formulate a person-centred health plan. This plan is part of and will be up-loaded to the eHealth platform which also contains individual notes and information about stress, depression and anxiety. The plan will be the point of departure for the forthcoming dialogue at distance via the eHealth platform that the patient and the RN will have during the study period (6 months).

The eHealth support contains headings that may inspire the patient to make notes on "a good day" respectively "a bad day" and register daily health related status. The health plan contain three parts; 1. "My goal is to feel or be able to do". 2. "To be able to reach my goal I will." 3."Support I need to reach my goal". In the communication during the study period between the RN and patient, the personal health plan is discussed and any needs of reformulating the goals may be discussed. The overall goal is to help the patient to identify their own capabilities/resources such as a strong will, social relations etc. and formulate goals that help them increase their self-efficacy and to cope with their condition in daily life.

The RN presents the eHealth support for communication (computer, iPad, smart phone) and they agree on how they will be in contact thereafter. The RN invites the patient and activates their account where he/she can login via an individual user name and formulate, comment, evaluate or develop the health plan. Access to the diary will be password protected. The RN can see the patient´s account and make comments. The patient can add or delete staff or private persons that have access to the account, and the patient can also limit the access for each user invited.

ELIGIBILITY:
Inclusion Criteria:

• Men and women fulfilling criteria for any of the following diagnoses: stress, depression or anxiety and on sick leave since ≤30 days

• Paid professional work, at least part time, during the last 9 months and willing to participate

Exclusion Criteria:

* Sick leave >14 days for any of the above mentioned diagnoses during the last 3 months.
* Severe impairment that prevents patient from using the eHealth support
* No registered address
* Not willing to participate
* Any severe disease with an expected survival <12 months
* Cognitive impairment
* Ongoing documented diagnosis of alcohol or drug abuse
* Other severe disease that can interfere with follow-up or if the intervention is assessed as a burden
* Patient participating in another conflicting randomized study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2018-02-14 (Actual); Primary Completion 2021-01-31 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Composite score of changes | baseline, 3, 6, 12, 18, 24 months
  A patient is classified as improved, deteriorated or unchanged:
  A patient is classified as improved if:
  at 6 months reduced sick leave and increased general self-efficacy by ≥ 5 units
  A patient is classified as deteriorated if:
  at 6 months increased sick leave or (if on full-time sick leave at inclusion reduced general self-efficacy by ≥ 5 units)
  Those who have neither deteriorated nor improved are considered unchanged

SECONDARY OUTCOMES:
Sick leave | baseline, 3, 6, 12, 18, 24 months
  Grade of sick leave
General self-efficacy scale | baseline, 3, 6, 12, 18, 24 months
  Questionnaire
Health-related quality of Life (EQ-5D) | baseline, 3, 6, 12, 18, 24 months
  Questionnaire
Hospital anxiety and depression scale (HADS) | baseline, 3, 6, 12, 18, 24 months
  Questionnaire
Symptom burden (Shirom-Melamed Burnout Measure) | baseline, 3, 6, 12, 18, 24 months
  Questionnaire
Perceived stress scale (PSS) | baseline, 3, 6, 12, 18, 24 months
  Questionnaire
Self-rated burnout syndrome (s-UMS) | baseline, 3, 6, 12, 18, 24 months
  Questionnaire
Health care utilization | 3, 6, 12, 18, 24 months
  Health care utilization
Incremental cost-utility ratios | 3, 6, 12, 18, 24 months
  Incremental cost-utility ratios
Multidimensional fatigue symptom inventory (MFI-20) | 3, 6, 12, 18, 24 months
  Questionnaire
Sheehan disability scale (SDS) | 3, 6, 12, 18, 24 months
  Questionnaire
Self-efficacy (self-care) | 3, 6, 12, 18, 24 months
  Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Fors, PhD, Principal Investigator — Institute of health and care sciences, Centre for person-centred care (GPCC)
Locations (1):
- Primary health care, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Alsen S, Cederberg M, Fors A. A person-centred care intervention provided via eHealth to reduce fatigue in patients with common mental disorders - secondary outcome analysis from a randomized controlled trial. Scand J Prim Health Care. 2025 Jul 24:1-10. doi: 10.1080/02813432.2025.2533997. Online ahead of print. PMID 40702943
- [Derived] Cederberg M, Barenfeld E, Ali L, Ekman I, Goulding A, Fors A. A lowered threshold to partnerships: a mixed methods process evaluation of participants' experiences of a person-centred eHealth intervention. BMC Health Serv Res. 2023 Nov 2;23(1):1193. doi: 10.1186/s12913-023-10190-7. PMID 37919705
- [Derived] Alsen S, Hadzibajramovic E, Jonsdottir IH, Ali L, Fors A. Effectiveness of a person-centred eHealth intervention in reducing symptoms of burnout in patients with common mental disorders - secondary outcome analysis of a randomized controlled trial. BMC Prim Care. 2023 Oct 19;24(1):210. doi: 10.1186/s12875-023-02172-9. PMID 37858032
- [Derived] Cederberg M, Alsen S, Ali L, Ekman I, Glise K, Jonsdottir IH, Gyllensten H, Swedberg K, Fors A. Effects of a Person-Centered eHealth Intervention for Patients on Sick Leave Due to Common Mental Disorders (PROMISE Study): Open Randomized Controlled Trial. JMIR Ment Health. 2022 Mar 15;9(3):e30966. doi: 10.2196/30966. PMID 35289756
- [Derived] Cederberg M, Ali L, Ekman I, Glise K, Jonsdottir IH, Gyllensten H, Swedberg K, Fors A. Person-centred eHealth intervention for patients on sick leave due to common mental disorders: study protocol of a randomised controlled trial and process evaluation (PROMISE). BMJ Open. 2020 Sep 1;10(9):e037515. doi: 10.1136/bmjopen-2020-037515. PMID 32873675